CLINICAL TRIAL: NCT05429216
Title: Modified Cap-assisted Endoscopic Mucosal Resection and Endoscopic Submucosal Dissection for Small Rectal Neuroendocrine Tumors Less Than 1 cm: a Muticenter Randomized Noninferiority Trial
Brief Title: Endoscopic Resection for Small Rectal Neuroendocrine Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-206
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-05

CONDITIONS: Rectal Neuroendocrine Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mEMR-C group (Experimental): In mEMR-C group, enrolled patients will receive modified EMR-C without submucosal injection.
  Interventions: Procedure: mEMR-C procedure
- ESD group (Active Comparator): In ESD group, enrolled patients will receive the standard treatment modality of ESD to remove the rectal NET
  Interventions: Procedure: ESD procedure

INTERVENTIONS:
Procedure: mEMR-C procedure — A transparent cap with an inner groove (MH-593; Olympus, Tokyo, Japan) was attached to the forward-viewing colonoscope. After the endoscope was inserted into the rectum, a crescent-shaped electrosurgical snare was passed through the sheath and looped along the inner groove of the cap. Submucosal injections were not required in this method. The tumor was suctioned into the cap and grasped by tightening the snare. After confirming the appropriate snare placement, both the tumor and overlying mucosa were resected using electric cautery (Endocut Q, effect 2, VIO 200D; ERBE, Tübingen, Germany), and the resected tumor was sent for pathological examination. Endoscopic examination was repeated without a transparent cap to evaluate the wound carefully in cases of perforation or bleeding and to ensure the absence of residual tumor tissues. If there was spurting or active bleeding, hot forceps were used to stop the bleeding.
  Arms: mEMR-C group
Procedure: ESD procedure — ESD was performed as the standard procedure and has been widely described and used. First, dots were marked approximately 5 mm from the periphery of the lesion using coagulation. Subsequently, a diluted sodium hyaluronate solution with indigo carmine dye was injected submucosally. Mucosal incision and submucosal dissection were performed using a T-Type ESD Knife (Micro-Tech, Nanjing, China) or Dual-knife (Olympus Medical, Tokyo, Japan). After resection was completed, all visible vessels on the artificial wound were thoroughly coagulated to prevent postoperative bleeding.
  Arms: ESD group

SUMMARY:
In previous single center study, both modified cap-assisted endoscopic mucosal resection (mEMR-C) and endoscopic submucosal dissection (ESD) were reported to be effective for the treatment of small rectal neuroendocrine tumors (NETs) and mEMR-C was inferior to ESD for the treatment of small rectal NETs (≤10 mm), as it has shorter operation times and lower hospitalization costs. However, a multicenter randomized controlled trial is needed to prove the universality and generality of these findings.

DETAILED DESCRIPTION:
Investigators aimed to conduct a muticenter randomized controlled trial to compare mEMR-C with ESD for the treatment of small rectal neuroendocrine tumors (NETs) in six tertiary hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years;
2. With a high suspicion or evidence of rectal NET assessed using EUS or colonoscopy;
3. With tumor size ≤10 mm assessed by colonoscopy;
4. Plan to receive mEMR-C or ESD treatment and provide written informed consent;

Exclusion Criteria:

1. Unable to tolerate ESD or MEMR-C as assessed by the research team of each center;
2. Complicated with serious diseases such as malignant tumor, which may lead to shorter life expectancy, the research team considers that it is not suitable for inclusion in the study after comprehensive evaluation;
3. Rectal NET with lymph node metastasis or distant metastasis;
4. Received resection of rectal neuroendocrine tumor by other surgical procedures;
5. Multiple rectal neuroendocrine tumors;
6. Vulnerable groups such as pregnant women or patients with mental disorders;
7. Poor compliance, unable to cooperate with treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
histological complete resection | within 14 days after procedure
  complete single-piece (en bloc) resection of the targeted lesion with horizontal and vertical free margins.

SECONDARY OUTCOMES:
success rate of operation | intraoperative
  the proportion of patients whose tumors were successfully resected in each group
en bloc resection | intraoperative
  complete single resection of the targeted lesion, irrespective of whether the basal and lateral tumor margins were infiltrated or undetermined
operation time | intraoperative
  the time required to complete the procedure, was taken from the installation of the snare in the mEMR-C or the first submucosal injection in ESD to the end of complete resection of the targeted area or a failure or complication of the procedure which required discontinuation
complications | within 14 days after procedure
  perforation or hemorrhage during or after operation.
length of stay | within 14 days after procedure
  calculated from the day of admission to day of discharge
hospitalization cost | within 14 days after procedure
  represent the hospital's costs of being hospitalized
operation cost | within 14 days after procedure
  the cost of mEMR-C or ESD procedures, except the cost of other endoscopic procedures
histopathologic grade | within 14 days after procedure
  NET grade 1, NET grade 2, NET grade 3, and NEC